CLINICAL TRIAL: NCT04142645
Title: Pilot Study of the OptiMEDs Intervention: a Complex Intervention for Multidisciplinary Medication Review (Including Nurses, Pharmacists, and Physicians) in Nursing Homes, With ICT-support for the Evaluation of the Appropriateness of Prescribing and for Side-effect Monitoring
Brief Title: OptiMEDs Pilot Study
Acronym: OptiMEDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B670201940251
Record Dates: First submitted 2019-09-30; First posted 2019-10-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Medication Review; Nursing Home Resident; Nursing Home
Keywords: Medication Reconciliation; Aged

STUDY DESIGN:
Intervention Model Description: A pragmatic cluster-randomized trial with the inclusion of two NHs where the feasibility and acceptability of the OptiMEDs intervention will be tested and one NH where the standard of care will be registered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group (i.e. all eligible and consented residents of 2 NHs) will receive the OptiMEDs intervention: the combination of an electronic decision support tool (for the appraisal of potentially inappropriate medication use, anticholinergic use, or medications that can be de-prescribed in view of limited life expectancy) with focused nurse observations (using a list of potential medication-related symptoms based on the individual medication chart of the nursing home residents), that will serve as the basis during a multidisciplinary medication review with the input of GPs, trained community pharmacists and nurses.
  Interventions: Device: OptiMEDs
- Control (No Intervention): The control group (i.e. all eligible and consented residents of one control NH) will receive usual care .

INTERVENTIONS:
Device: OptiMEDs — The OptiMEDs intervention is a multi-faceted intervention combining:
  1. an ICT platform:
     * automatic and secure capture of individual prescribing information from the electronic medication administration records in the nursing home
     * a tool for structured nurse observations of side effects, derived from the existing Pharmanurse application (20) (used to list potential medication side effects, based on the individual medication chart of the nursing home residents) to support monitoring of medication safety by nurses.
     * an electronic decision support tool for the appraisal of potentially inappropriate medication (explicit criteria of misuse and underused of medication, based on existing lists of explicit criteria (PIMs)), use of medication with anticholinergic properties and medication inappropriate in view of the limited life expectancy.
  2. a multidisciplinary medication review with the input of GPs, trained community-pharmacists and nurses.
  Arms: Intervention

SUMMARY:
Pilot study of the OptiMEDs intervention: a complex intervention for multidisciplinary medication review (including nurses, pharmacists, and physicians) in nursing homes (NH), with ICT-support for the evaluation of the appropriateness of prescribing and for side-effect monitoring.

DETAILED DESCRIPTION:
The interest in improving the pharmacotherapy of older adults in nursing homes is growing. The OptiMEDs interventions intends to support the decision of GPs regarding the pharmacotherapy of older adults through the combination of an electronic decision support tool (for the appraisal of potentially inappropriate medication use, anticholinergic use, or medications that can be de-prescribed in view of limited life expectancy) with focussed nurse observations (guided by a list of potential medication symptoms based on the individual medication chart of the resident), that will serve as the basis for a multidisciplinary medication review with the input of the GP, community pharmacist and nurse.

The aim of the OptiMEDs intervention is to obtain a more appropriate, safer, and more cost-effective pharmacotherapy in nursing home residents (e.g. less medication-related symptoms, less potentially inappropriate prescribing, a better quality of life, less hospitalisations, health care usage, or mortality)

Before investigating the effectiveness of the OptiMEDs intervention in a large pragmatic clinical trial comparing results of the intervention with standard of care, a pilot study will be undertaken. The aim of the pilot study is to test the feasibility and acceptability of all components of the OptiMEDs interventions in 3 nursing homes in Flanders, Belgium.

ELIGIBILITY:
Inclusion criteria for nursing homes:

* located in East Flanders
* size: > 100 beds
* mixed population of high care dependent and low care-dependent residents with and without dementia
* software of Care Solutions or Farmad is used for electronic handling of the medication chart
* the NH management as well as the responsible CRA and the community pharmacist who delivers the medication in the NH give their written agreement to participate

Inclusion criteria for residents:

All residents of all wards of the participating nursing homes will be considered for inclusion if they meet the following inclusion criteria:

* aged 65 years or older
* mentally fit as well as cognitive impaired NH residents will be included after Informed Consent given by the resident (mentally capable residents) or his representative (cognitive impaired residents, defined as a sumscore of 6 or more on the KATZ items of disorientation in time and place).

Exclusion criteria for residents

Residents will not be considered for inclusion if:

* they have a limited life-expectancy (less than 3 months, as judged and documented by the treating GP)
* they are residing in a short-stay / revalidation bed
* GP refused to have his NH residents included in this pilot

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Software/user problems | 6 months
  monthly number of interventions for software/user problems (n)
functionality problems | 6 months
  Number of functionality problems (n)
workload | 6 months
  Timing of workload for nurses & pharmacists regarding the use of OptiMEDs (time)
medication chart review | 6 months
  duration of a medication chart review by GP and nurse (time)
practical problems | 6 months
  listing of practical problems for organizing the medication chart review
GPs that refuse | 6 months
  number of GPs that refuse to participate / accept to participate (n)
non-consenting eligible residents (n) | 6 months
  Number of non-consenting eligible residents legally capable to give consent (n)
Non-consenting proxies for eligible residents (n) | 6 months
  Number of non-consenting proxies for eligible residents legally not capable to give consent
Optimeds completion | 6 months
  Number of symptom observations and medication reviews completed (on time) (n)

SECONDARY OUTCOMES:
number of medications | 4 months
  number of medications (n)
number of anticholinergics | 4 months
  number of anticholinergics (n)
number of candidates for de-prescribing | 4 months
  number of candidates for de-prescribing (n)
patient-related pain | 4 months
  Score; In patients with dementia: nurse-observation using PAIN-AD scale (0 - 10, 10 = worst pain), patients without dementia: Pain VAS scale (0 - 10, 10 = worst pain)
patient-related alertness | 4 months
  patient-related alertness (score); nurse-observation using VAS scale (1 - 6, 1 = being alert)
patient-related QOL | 4 months
  patient-related QOL (score and/or profile); EQ-5D-5L; 5 dimensions (mobility / self-care / usual activities / pain or discomfort / anxiety or depression) and 5 levels (no / slight / moderate / severe / extreme problems).
patient-related falls | 4 months
  patient-related falls (n)
Number of Consultations | 4 months
  Number of Consultations (n)
Number of Hospitalization | 4 months
  Number of Hospitalization (n)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Christiaens, PhD, MD, Principal Investigator — Faculty of Medicine and Health Sciences
Locations (3):
- Belgium (3):
  - WZC Sint-Jozef Deinze, Deinze, Oost-Vlaanderen
  - WZC Sint-Jozef Gent, Ghent, Oost-Vlaanderen
  - WZC Liberteyt, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Almeida Mello J, Van Durme T, Macq J, Declercq A. Interventions to delay institutionalization of frail older persons: design of a longitudinal study in the home care setting. BMC Public Health. 2012 Aug 6;12:615. doi: 10.1186/1471-2458-12-615. PMID 22867442
- [Background] Azermai M, Elseviers M, Petrovic M, Van Bortel L, Vander Stichele R. Geriatric drug utilisation of psychotropics in Belgian nursing homes. Hum Psychopharmacol. 2011 Jan;26(1):12-20. doi: 10.1002/hup.1160. PMID 21394786
- [Background] Mann E, Kopke S, Haastert B, Pitkala K, Meyer G. Psychotropic medication use among nursing home residents in Austria: a cross-sectional study. BMC Geriatr. 2009 May 21;9:18. doi: 10.1186/1471-2318-9-18. PMID 19460135
- [Background] Turnheim K. When drug therapy gets old: pharmacokinetics and pharmacodynamics in the elderly. Exp Gerontol. 2003 Aug;38(8):843-53. doi: 10.1016/s0531-5565(03)00133-5. PMID 12915206
- [Background] Klotz U. Pharmacokinetics and drug metabolism in the elderly. Drug Metab Rev. 2009;41(2):67-76. doi: 10.1080/03602530902722679. PMID 19514965
- [Background] Basger BJ, Moles RJ, Chen TF. Application of drug-related problem (DRP) classification systems: a review of the literature. Eur J Clin Pharmacol. 2014 Jul;70(7):799-815. doi: 10.1007/s00228-014-1686-x. Epub 2014 May 2. PMID 24789053
- [Background] Shenoy P, Harugeri A. Elderly patients' participation in clinical trials. Perspect Clin Res. 2015 Oct-Dec;6(4):184-9. doi: 10.4103/2229-3485.167099. PMID 26623388
- [Background] Anrys P, Strauven G, Boland B, Dalleur O, Declercq A, Degryse JM, De Lepeleire J, Henrard S, Lacour V, Simoens S, Speybroeck N, Vanhaecht K, Spinewine A, Foulon V. Collaborative approach to Optimise MEdication use for Older people in Nursing homes (COME-ON): study protocol of a cluster controlled trial. Implement Sci. 2016 Mar 11;11:35. doi: 10.1186/s13012-016-0394-6. PMID 26968520
- [Background] Azermai M, Wauters M, De Meester D, Renson L, Pauwels D, Peeters L, Warie H, Petrovic M. A quality improvement initiative on the use of psychotropic drugs in nursing homes in Flanders. Acta Clin Belg. 2017 Jun;72(3):163-171. doi: 10.1080/17843286.2017.1287230. Epub 2017 Feb 16. PMID 28206874
- [Background] Ivanova I, Elseviers M, Wauters M, Christiaens T, Vander Stichele R. European repository of explicit criteria of potentially inappropriate medications in old age. Geriatr Gerontol Int. 2018 Aug;18(8):1293-1297. doi: 10.1111/ggi.13331. Epub 2018 Apr 17. PMID 29665270
- [Background] Robertson J, Walkom E, Pearson SA, Hains I, Williamsone M, Newby D. The impact of pharmacy computerised clinical decision support on prescribing, clinical and patient outcomes: a systematic review of the literature. Int J Pharm Pract. 2010 Apr;18(2):69-87. PMID 20441116
- [Background] Lavan AH, Gallagher PF, O'Mahony D. Methods to reduce prescribing errors in elderly patients with multimorbidity. Clin Interv Aging. 2016 Jun 23;11:857-66. doi: 10.2147/CIA.S80280. eCollection 2016. PMID 27382268
- [Background] Forsetlund L, Eike MC, Gjerberg E, Vist GE. Effect of interventions to reduce potentially inappropriate use of drugs in nursing homes: a systematic review of randomised controlled trials. BMC Geriatr. 2011 Apr 17;11:16. doi: 10.1186/1471-2318-11-16. PMID 21496345
- [Background] Alldred DP, Raynor DK, Hughes C, Barber N, Chen TF, Spoor P. Interventions to optimise prescribing for older people in care homes. Cochrane Database Syst Rev. 2013 Feb 28;(2):CD009095. doi: 10.1002/14651858.CD009095.pub2. PMID 23450597
- [Background] Majumdar SR, Soumerai SB. Why most interventions to improve physician prescribing do not seem to work. CMAJ. 2003 Jul 8;169(1):30-1. No abstract available. PMID 12847036
- [Background] Grimshaw JM, Shirran L, Thomas R, Mowatt G, Fraser C, Bero L, Grilli R, Harvey E, Oxman A, O'Brien MA. Changing provider behavior: an overview of systematic reviews of interventions. Med Care. 2001 Aug;39(8 Suppl 2):II2-45. PMID 11583120
- [Background] Patterson SM, Hughes C, Kerse N, Cardwell CR, Bradley MC. Interventions to improve the appropriate use of polypharmacy for older people. Cochrane Database Syst Rev. 2012 May 16;(5):CD008165. doi: 10.1002/14651858.CD008165.pub2. PMID 22592727
- [Background] Huiskes VJ, Burger DM, van den Ende CH, van den Bemt BJ. Effectiveness of medication review: a systematic review and meta-analysis of randomized controlled trials. BMC Fam Pract. 2017 Jan 17;18(1):5. doi: 10.1186/s12875-016-0577-x. PMID 28095780
- [Background] Dilles T, Vander Stichele RH, Van Bortel LM, Elseviers MM. The development and test of an intervention to improve ADR screening in nursing homes. J Am Med Dir Assoc. 2013 May;14(5):379.e1-6. doi: 10.1016/j.jamda.2013.02.011. Epub 2013 Apr 2. PMID 23557831
- [Background] Wouters H, Scheper J, Koning H, Brouwer C, Twisk JW, van der Meer H, Boersma F, Zuidema SU, Taxis K. Discontinuing Inappropriate Medication Use in Nursing Home Residents: A Cluster Randomized Controlled Trial. Ann Intern Med. 2017 Nov 7;167(9):609-617. doi: 10.7326/M16-2729. Epub 2017 Oct 10. PMID 29052691
- [Background] Wauters M, Elseviers M, Vaes B, Degryse J, Dalleur O, Vander Stichele R, Christiaens T, Azermai M. Too many, too few, or too unsafe? Impact of inappropriate prescribing on mortality, and hospitalization in a cohort of community-dwelling oldest old. Br J Clin Pharmacol. 2016 Nov;82(5):1382-1392. doi: 10.1111/bcp.13055. Epub 2016 Aug 3. PMID 27426227
- [Background] Wauters M, Elseviers M, Azermai M, Vander Stichele R. Availability and actual use in the Belgian market of potentially inappropriate medications (PIMs) from the EU(7)-PIM list. Eur J Clin Pharmacol. 2016 Feb;72(2):243-5. doi: 10.1007/s00228-015-1947-3. Epub 2015 Sep 26. No abstract available. PMID 26407685
- [Background] Duran CE, Azermai M, Vander Stichele RH. Systematic review of anticholinergic risk scales in older adults. Eur J Clin Pharmacol. 2013 Jul;69(7):1485-96. doi: 10.1007/s00228-013-1499-3. Epub 2013 Mar 26. PMID 23529548
- [Background] Klamer TT, Wauters M, Azermai M, Duran C, Christiaens T, Elseviers M, Vander Stichele R. A Novel Scale Linking Potency and Dosage to Estimate Anticholinergic Exposure in Older Adults: the Muscarinic Acetylcholinergic Receptor ANTagonist Exposure Scale. Basic Clin Pharmacol Toxicol. 2017 Jun;120(6):582-590. doi: 10.1111/bcpt.12699. Epub 2017 Jan 16. PMID 28090742
- [Background] Wauters M, Klamer T, Elseviers M, Vaes B, Dalleur O, Degryse J, Duran C, Christiaens T, Azermai M, Vander Stichele R. Anticholinergic Exposure in a Cohort of Adults Aged 80 years and Over: Associations of the MARANTE Scale with Mortality and Hospitalization. Basic Clin Pharmacol Toxicol. 2017 Jun;120(6):591-600. doi: 10.1111/bcpt.12744. Epub 2017 Apr 6. PMID 27995743
- [Background] Morin L, Laroche ML, Vetrano DL, Fastbom J, Johnell K. Adequate, questionable, and inadequate drug prescribing for older adults at the end of life: a European expert consensus. Eur J Clin Pharmacol. 2018 Oct;74(10):1333-1342. doi: 10.1007/s00228-018-2507-4. Epub 2018 Jun 23. PMID 29934849
- [Background] Poudel A, Yates P, Rowett D, Nissen LM. Use of Preventive Medication in Patients With Limited Life Expectancy: A Systematic Review. J Pain Symptom Manage. 2017 Jun;53(6):1097-1110.e1. doi: 10.1016/j.jpainsymman.2016.12.350. Epub 2017 Feb 9. PMID 28192226
- [Background] Todd A, Husband A, Andrew I, Pearson SA, Lindsey L, Holmes H. Inappropriate prescribing of preventative medication in patients with life-limiting illness: a systematic review. BMJ Support Palliat Care. 2017 Jun;7(2):113-121. doi: 10.1136/bmjspcare-2015-000941. Epub 2016 Jan 5. PMID 26733578
- [Background] Warden V, Hurley AC, Volicer L. Development and psychometric evaluation of the Pain Assessment in Advanced Dementia (PAINAD) scale. J Am Med Dir Assoc. 2003 Jan-Feb;4(1):9-15. doi: 10.1097/01.JAM.0000043422.31640.F7. PMID 12807591
- [Background] Ivanova I, Wauters M, Stichele RV, Christiaens T, De Wolf J, Dilles T, Elseviers M. Medication use in a cohort of newly admitted nursing home residents (Ageing@NH) in relation to evolving physical and mental health. Arch Gerontol Geriatr. 2018 Mar-Apr;75:202-208. doi: 10.1016/j.archger.2018.01.005. Epub 2018 Jan 17. PMID 29353187
- [Derived] Wauters M, Elseviers M, Vander Stichele R, Dilles T, Thienpont G, Christiaens T. Efficacy, feasibility and acceptability of the OptiMEDs tool for multidisciplinary medication review in nursing homes. Arch Gerontol Geriatr. 2021 Jul-Aug;95:104391. doi: 10.1016/j.archger.2021.104391. Epub 2021 Mar 17. PMID 33819776